CLINICAL TRIAL: NCT04353882
Title: Evaluation of the Difference in Expression of the Mu Type 1 Opioid Receptor and of the Markers of Its Activation (Cyclic Adenosine Monophosphate and Protein Kinase A) in Colorectal Cancer. Case-control Study in Patients With Tumor Recurrence Versus Disease-free Patients at 5 Years.
Brief Title: Mu Opioid Receptor 1 Expression and Activation Patterns in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Principal Investigator of Anesthesiology, Hospital Universitario La Fe
Other Study IDs: MOROCCO-II
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Surgery for Stage II / III Primary Colorectal Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with tumor recurrence
  Interventions: Other: Assess the difference in MOR-1 expression between healthy and tumor tissue
- patients with-out tumor recurrence
  Interventions: Other: Assess the difference in MOR-1 expression between healthy and tumor tissue

INTERVENTIONS:
Other: Assess the difference in MOR-1 expression between healthy and tumor tissue — Assess the difference in the quantitative expression of MOR-1 (by means of RT-qPCR) between healthy tissue and tumor tissue, in patients with stage II and III colorectal cancer undergoing scheduled surgery.

SUMMARY:
Observational case-control study in a retrospective cohort of patients with stage II or III colorectal cancer undergoing scheduled surgery.

DETAILED DESCRIPTION:
Observational case-control study in a retrospective cohort of patients with stage II or III colorectal cancer undergoing scheduled surgery. Period January 2010-December 2014. Patients must have had at least 5 years of follow-up to define disease-free survival. From the cohort of patients previously studied in our center by immunohistochemistry, 31 we will select 10 cases with recurrence by random sampling and we will match 10 controls by leveling the propensity score (propensity score matching).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Colorectal surgery scheduled between January 2010 - December 2014.
* Stage II or III colon or rectum neoplasm (T3 / T4 N + M0).

Exclusion Criteria:

* Neoplasia of colon or rectum in Stage I or Stage IV.
* Non-oncological colorectal surgery.
* Urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled colorectal surgery for stage II and III primary colorectal cancer during the period 01/01/2010 and 12/31/2014.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
MOR-1 expression by polymerase chain reaction (RT-qPCR) in tumor tissue and adjacent healthy tissue. | Day 1

SECONDARY OUTCOMES:
Cancer-free survival 5 years after surgery (disease-free survival-DFS). | Day 1
Degree of MOR-1 activation measured by immunohistochemistry through cAMP and PKA levels. | Day 1
MOR-1 expression by immunohistochemistry in tumor tissue and adjacent healthy tissue. | Day 1

OTHER OUTCOMES:
Use of halogenated vs intravenous hypnotic agent | Day 1
Carcinoembryonic antigen | Day 1
Cancer antigen | Day 1
Neoadjuvant or adjuvant chemotherapy or radiation therapy | Day 1
Surgery time | Day 1
Surgery date | Day 1
Hospital discharge | Day 1
Surgery complications | Day 1
Type of surgery | Day 1
ASA test | Day 1
Concomitant Diseases | Day 1